CLINICAL TRIAL: NCT04755257
Title: Development of the Muscle Architecture Based Isokinetic Strength Assessment Position for Shoulder Rotator Muscles
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, caglar soylu, Çağlar Soylu (Principal Investigator), Ankara Yildirim Beyazıt University
Other Study IDs: 2019-367
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Muscle Architecture; Shoulder; Isokinetic; Rotator Muscle
Keywords: Muscle Architecture; Shoulder; Isokinetic; Rotator muscle

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Isokinetic test — Using IsoMed 2000 device (D. & R. Ferstl GmbH, Hemau, Germany) we conducted the isokinetic test of concentric (CON) and eccentric (ECC) shoulder internal (IR) and external (ER) strength at the angular velocity of 60˚/s in both Method I (scapular position) and Method II (25⁰ Abd and 20⁰ ER). There were seven days between the testing sessions, and both tests were conducted at the same time of day. The same examiner with experience in performing isokinetic testing with IsoMed 2000 tested all subjects in both testing sessions.

SUMMARY:
Today, the most commonly used position is the seated position with 45° of shoulder abduction (Abd) in the scapular plane, known as the most functional isokinetic assessment of shoulder-rotator strength (1). However, considering the architectural feature of the rotator muscles, a position where the maximum sarcomere length is obtained, in which the maximum muscle strength is produced, has not been investigated. Ward et al. showed that the shoulder position, in which the sarcomere length of the muscles was between 2.0 - 2.6 µm, was 25⁰ Abd and 20⁰ external rotation (ER) as a result of their study on the rotator cuff muscles architecture (2). The test position selected in isokinetic measurements is the main factor for outcome measurements and the repeatability of the measurements directly depends on the selected position (3). This study was planned to investigate the effects of the position where the shoulder is at 25⁰ Abd and 20⁰ ER to develop the most suitable isokinetic strength evaluation position based on muscle architecture for shoulder rotator muscles.Using IsoMed 2000 device (D. & R. Ferstl GmbH, Hemau, Germany) we conducted the isokinetic test of concentric (CON) and eccentric (ECC) shoulder internal (IR) and external (ER) strength at the angular velocity of 60˚/s in both Method I (scapular position) and Method II (25⁰ Abd and 20⁰ ER). There were seven days between the testing sessions, and both tests were conducted at the same time of day. The same examiner with experience in performing isokinetic testing with IsoMed 2000 tested all subjects in both testing sessions

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-25
* Body mass index (BMI) being between 18.5-24.9 kg / m 2
* Volunteering to participate in the study
* Having the skills to do the tests and exercises to be applied

Exclusion Criteria:

* Having a history of upper extremity injury within the past year
* Having a sensory problem that prevents participation in the study
* Have any musculoskeletal, neurological, respiratory, or cardiovascular risk factors that limit exercise
* Having a history of malignant disease

Ages: 18 Years to 25 Years | Sex: Male
Age Groups: Adult
Gender Based: Yes — healthy male subjects
Study Population: healthy male subjects
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
concentric shoulder internal rotation peak torque and peak torque/weight at the angular velocity of 60˚/s in Method I (scapular position) | Six month
  concentric shoulder internal rotation peak torque and peak torque/weight at the angular velocity of 60˚/s in Method I (scapular position)
concentric shoulder external rotation peak torque and peak torque/weight at the angular velocity of 60˚/s in Method I (scapular position) | Six month
  concentric shoulder external rotation peak torque and peak torque/weight at the angular velocity of 60˚/s in Method I (scapular position)
concentric shoulder internal rotation peak torque and peak torque/weight at the angular velocity of 60˚/s in Method II (25⁰ Abd and 20⁰ ER) | Six month
  concentric shoulder internal rotation peak torque and peak torque/weight at the angular velocity of 60˚/s in Method II (25⁰ Abd and 20⁰ ER)
concentric shoulder external rotation peak torque and peak torque/weight at the angular velocity of 60˚/s in Method II (25⁰ Abd and 20⁰ ER) | Six month
  concentric shoulder external rotation peak torque and peak torque/weight at the angular velocity of 60˚/s in Method II (25⁰ Abd and 20⁰ ER)
eccentric shoulder internal rotation peak torque and peak torque/weight at the angular velocity of 60˚/s in Method I (scapular position) | Six month
  eccentric shoulder internal rotation peak torque and peak torque/weight at the angular velocity of 60˚/s in Method I (scapular position)
eccentric shoulder external rotation peak torque and peak torque/weight at the angular velocity of 60˚/s in Method I (scapular position) | Six month
  eccentric shoulder external rotation peak torque and peak torque/weight at the angular velocity of 60˚/s in Method I (scapular position)
eccentric shoulder internal rotation peak torque and peak torque/weight at the angular velocity of 60˚/s in Method II (25⁰ Abd and 20⁰ ER) | Six month
  eccentric shoulder internal rotation peak torque and peak torque/weight at the angular velocity of 60˚/s in Method II (25⁰ Abd and 20⁰ ER)
eccentric shoulder external rotation peak torque and peak torque/weight at the angular velocity of 60˚/s in Method II (25⁰ Abd and 20⁰ ER) | Six month
  eccentric shoulder external rotation peak torque and peak torque/weight at the angular velocity of 60˚/s in Method II (25⁰ Abd and 20⁰ ER)

CONTACTS AND LOCATIONS:
Overall Officials: Caglar Soylu, PhD, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yıldırım Beyazıt University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Etlik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No